CLINICAL TRIAL: NCT02753114
Title: Prehospital Analgesia With Intra-Nasal Ketamine
Acronym: PAIN-K
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: British Columbia Emergency Health Services (Unknown)
Responsible Party: Principal Investigator, Gary Andolfatto, Assistant Professor, University of British Columbia Department of Emergency Medicine, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H16-00554
Record Dates: First submitted 2016-04-16; First posted 2016-04-27 (Estimated); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Pain; Acute Pain
Keywords: Ketamine; Intranasal; Emergency Medical Services; Pain; Analgesia
MeSH Terms: conditions — Pain; Acute Pain; Agnosia | interventions — Ketamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intranasal Ketamine (Experimental): Ketamine dosing will be weight-based as follows: 30mg of IN ketamine for patients weighing 50 kg or less; 50 mg of IN ketamine for patients weighing 50 kg to 100 kg; and 75 mg of IN ketamine for patients weighing greater than 100 kg (i.e. 0.5 mg/kg to 1.0 mg/kg of intranasal ketamine). Syringes containing ketamine will be prepared from the intravenous formulation of Ketamine (50 mg / ml) solution (Sandoz; DIN 02246796) and stored in pre-filled 5 ml syringes. Ketamine will be administered to patients through a mucosal atomization device. One-half of the pre-specified volume will be administered into each nare. No repeat doses will be administered.
  Interventions: Drug: Ketamine
- Placebo (Placebo Comparator): Syringes containing normal saline will be prepared such that the volume of normal saline in 5 ml syringes matches that of the ketamine for each of the weight based groups previously specified in the Treatment Arm Description. Syringes containing normal saline will also be labeled "Study Drug". The normal saline will also be administered to patients through a mucosal atomization device. One-half of the pre-specified volume will be administered into each nare. No repeat doses of placebo will be administered.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Ketamine — Intranasal Ketamine administered via mucosal atomization device at 0.5 - 1 mg / kg IN.
  Other Names: Sandoz DIN 02246796; Ketalar
  Arms: Intranasal Ketamine
Drug: Normal Saline — Intranasal Normal Saline administered via mucosal atomization device.
  Other Names: Saline placebo
  Arms: Placebo

SUMMARY:
Acute painful conditions make-up a large proportion of pre-hospital transports in British Columbia (BC) yet Basic Life Support (BLS) paramedics have limited options to provide analgesia and therefore adequate and timely pain relief is often significantly delayed.

Inhaled nitrous oxide is commonly used as a pre-hospital analgesic and is considered "usual care" for pre-hospital providers in BC, but its utility in severe pain is uncertain. Moreover, nitrous oxide is limited in its effectiveness by a short duration of action, nausea, vomiting, and the necessity for patient cooperation.

IN Ketamine has been shown to provide rapid, easily-administered, and well-tolerated analgesia in many settings. The investigators believe that the addition of IN ketamine to usual care with nitrous oxide inhalation for adults experiencing moderate to severe intensity acute pain in the pre-hospital setting will result in improved pain severity, improved patient-reported comfort, and improved patient satisfaction.

DETAILED DESCRIPTION:
Purpose:

The purpose of this study is to see whether intra-nasal (IN) Ketamine (50 mg / ml) solution (Sandoz; Drug Identification Number (DIN) 02246796) administered via mucosal atomization device (LMA MAD300 Nasal TM; Wolfe Tory Medical Inc., San Diego, CA), in addition to usual care with nitrous oxide inhalation, to pre-hospital patients being transported by British Columbia Emergency Health Services (BC EHS) Basic Life Support (BLS) paramedics with moderate to severe pain (pain > 5/10 on a validated numerical rating scale or NRS) will improve pain relative to usual care plus placebo.

Hypothesis:

It is hypothesized that the addition of IN ketamine to usual care with nitrous oxide inhalation for adults experiencing moderate to severe intensity acute pain in the pre-hospital setting will result in a greater proportion of patients experiencing a 2-point or more reduction in verbal numerical rating scale (VNRS) pain score within 30 minutes, as well as improved patient-reported comfort, reduced nitrous oxide requirements, and improved patient and provider satisfaction compared to usual care alone.

Background:

Acute painful conditions make-up a large proportion of pre-hospital transports yet BLS paramedics have limited options to provide analgesia, and therefore, adequate and timely pain relief is often significantly delayed. Inhaled nitrous oxide is commonly used as a pre-hospital analgesic and is considered "usual care" for BLS pre-hospital providers. Nitrous oxide has been shown to be effective for analgesia in patients with moderate pain but its utility in severe pain is uncertain. No alternative treatments exist for BLS providers in the pre-hospital setting. Intra-nasal ketamine is a safe, well-tolerated means of providing analgesia and has been proven to work in the pre-hospital setting without the need for cardio-respiratory monitoring.

Objectives:

The objective of this study is to collect pilot data to compare the addition of intranasal Ketamine or an intranasal placebo in terms of efficacy and effectiveness in patients receiving usual care with nitrous oxide for moderate to severe pain.

Secondary objectives will be to assess subjective improvement in pain, effect on nitrous oxide requirements, incidence of adverse effects, patient and provider satisfaction, and study recruitment potential. These data will inform future large-scale trial designs and will be used to validate a proposed 7-point patient-reported pain improvement scale.

Research Methods:

This will be a randomized double-blind pilot trial conducted in the pre-hospital setting in the lower mainland. The pilot series will constitute 40 patients (20 per group). The sample size for a larger randomized controlled trial will then be calculated using the effect size and variance of the accrued data.

Statistical Analysis:

A statistician will be contracted to independently oversee the analysis of study results. The intention-to-treat principal will be used to analyze all data. Data will be analyzed using descriptive statistics. Categorical data will be presented as frequency and percentage frequency of occurrence. Continuous data will be presented as medians with ranges and interquartile ranges (IQRs). Adverse effects will be described as frequency of occurrence with 95% confidence intervals. A p-value of 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have an acute painful condition, as determined by the Emergency Health Services attendant
* A pain score of 5 or greater (signifying moderate or severe pain)
* Desire for analgesia when queried.

Exclusion Criteria:

* Less than 18 years of age.
* Previous hypersensitivity, intolerance or allergy to ketamine
* Chest pain
* Altered mental status
* Inability self-report pain score
* Pregnancy
* Nasal occlusion
* Systolic Blood Pressure < 90 mm Hg
* Requiring immediate attention of the paramedic
* Ineligible to receive inhaled nitrous oxide as per BC EHS protocols

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2018-05-24 (Actual); Study Completion 2018-05-24 (Actual)

PRIMARY OUTCOMES:
Proportion experiencing 2-point or more pain score reduction at 30 minutes | 30 minutes.
  The proportion of patients experiencing a 2-point or more reduction in NRS pain score at 30 minutes.

SECONDARY OUTCOMES:
Proportion experiencing 2-point or more pain score reduction at 15 minutes | 15 minutes
  The proportion of patients experiencing a 2-point or more reduction in NRS pain score at 15 minutes.
The proportion of patients feeling "a lot better" or "moderately better" at 30 minutes post medication delivery or hospital at hospital arrival | 30 minutes
  The proportion of patients feeling "a lot better" or "moderately better" at 30 minutes post medication delivery or hospital at hospital arrival
The proportion of patients feeling "a lot better" or "moderately better" at 15 minutes. | 15 minutes
  The proportion of patients feeling "a lot better" or "moderately better" at 15 minutes.
The proportion of patients feeling "a lot better", "moderately better" or "a little better" at 15 minutes and at 30 minutes. | 15 minutes, 30 minutes
  The proportion of patients feeling "a lot better", "moderately better" or "a little better" at 15 minutes and at 30 minutes.
Adverse Events | Every 15 minutes until care transferred to Emergency Department
  Incidence of adverse events.
Patient Satisfaction | At 30 minutes post analgesia administration.
  Patient satisfaction with analgesia provided using a ten point numeric rating scale anchored with 0 = "not at all satisfied" and 10 = "completely satisfied" on hospital arrival.
Provider Satisfaction | At 30 minutes post analgesia administration.
  Paramedic satisfaction with analgesia provided using a ten point numeric rating scale anchored with 0 = "not at all satisfied" and 10 = "completely satisfied" on hospital arrival.
Median Nitrous Oxide Consumption | At 30 minutes post analgesia administration.
  Median nitrous oxide consumption in each group will be recorded and compared.
Median reduction in pain score at 15 minutes | 15 minutes
  Median reduction in NRS pain score at 15 minutes
Median reduction in pain score at 30 minutes | 30 minutes
  Median reduction in NRS pain score at 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Gary Andolfatto, Principal Investigator — University of British Columbia
Locations (1):
- British Columbia Emergency Health Services Station 249, Surrey, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Murphy A, McCoy S, O'Reilly K, Fogarty E, Dietz J, Crispino G, Wakai A, O'Sullivan R. A Prevalence and Management Study of Acute Pain in Children Attending Emergency Departments by Ambulance. Prehosp Emerg Care. 2016;20(1):52-8. doi: 10.3109/10903127.2015.1037478. Epub 2015 May 29. PMID 26024309
- [Background] McLean SA, Maio RF, Domeier RM. The epidemiology of pain in the prehospital setting. Prehosp Emerg Care. 2002 Oct-Dec;6(4):402-5. doi: 10.1080/10903120290938021. PMID 12385606
- [Background] Marinangeli F, Narducci C, Ursini ML, Paladini A, Pasqualucci A, Gatti A, Varrassi G. Acute pain and availability of analgesia in the prehospital emergency setting in Italy: a problem to be solved. Pain Pract. 2009 Jul-Aug;9(4):282-8. doi: 10.1111/j.1533-2500.2009.00277.x. Epub 2009 Mar 16. PMID 19490463
- [Background] Lord B, Cui J, Kelly AM. The impact of patient sex on paramedic pain management in the prehospital setting. Am J Emerg Med. 2009 Jun;27(5):525-9. doi: 10.1016/j.ajem.2008.04.003. PMID 19497456
- [Background] Jennings PA, Cameron P, Bernard S. Epidemiology of prehospital pain: an opportunity for improvement. Emerg Med J. 2011 Jun;28(6):530-1. doi: 10.1136/emj.2010.098954. Epub 2010 Aug 2. PMID 20679429
- [Background] Chambers JA, Guly HR. The need for better pre-hospital analgesia. Arch Emerg Med. 1993 Sep;10(3):187-92. doi: 10.1136/emj.10.3.187. PMID 8216592
- [Background] Ducasse JL, Siksik G, Durand-Bechu M, Couarraze S, Valle B, Lecoules N, Marco P, Lacombe T, Bounes V. Nitrous oxide for early analgesia in the emergency setting: a randomized, double-blind multicenter prehospital trial. Acad Emerg Med. 2013 Feb;20(2):178-84. doi: 10.1111/acem.12072. PMID 23406077
- [Background] Oglesbee S, Selde W. Nitrous oxide. New delivery of an old drug. JEMS. 2014 Apr;39(4):34-7. No abstract available. PMID 24779097
- [Background] Faddy SC, Garlick SR. A systematic review of the safety of analgesia with 50% nitrous oxide: can lay responders use analgesic gases in the prehospital setting? Emerg Med J. 2005 Dec;22(12):901-8. doi: 10.1136/emj.2004.020891. PMID 16299211
- [Background] Johansson J, Sjoberg J, Nordgren M, Sandstrom E, Sjoberg F, Zetterstrom H. Prehospital analgesia using nasal administration of S-ketamine--a case series. Scand J Trauma Resusc Emerg Med. 2013 May 14;21:38. doi: 10.1186/1757-7241-21-38. PMID 23672762
- [Background] Borland ML, Jacobs I, Geelhoed G. Intranasal fentanyl reduces acute pain in children in the emergency department: a safety and efficacy study. Emerg Med (Fremantle). 2002 Sep;14(3):275-80. doi: 10.1046/j.1442-2026.2002.00344.x. PMID 12487045
- [Background] Borland M, Jacobs I, King B, O'Brien D. A randomized controlled trial comparing intranasal fentanyl to intravenous morphine for managing acute pain in children in the emergency department. Ann Emerg Med. 2007 Mar;49(3):335-40. doi: 10.1016/j.annemergmed.2006.06.016. Epub 2006 Oct 25. PMID 17067720
- [Background] Borland ML, Clark LJ, Esson A. Comparative review of the clinical use of intranasal fentanyl versus morphine in a paediatric emergency department. Emerg Med Australas. 2008 Dec;20(6):515-20. doi: 10.1111/j.1742-6723.2008.01138.x. PMID 19125831
- [Background] Holdgate A, Cao A, Lo KM. The implementation of intranasal fentanyl for children in a mixed adult and pediatric emergency department reduces time to analgesic administration. Acad Emerg Med. 2010 Feb;17(2):214-7. doi: 10.1111/j.1553-2712.2009.00636.x. PMID 20070272
- [Background] Karlsen AP, Pedersen DM, Trautner S, Dahl JB, Hansen MS. Safety of intranasal fentanyl in the out-of-hospital setting: a prospective observational study. Ann Emerg Med. 2014 Jun;63(6):699-703. doi: 10.1016/j.annemergmed.2013.10.025. Epub 2013 Nov 22. PMID 24268523
- [Background] Jennings PA, Cameron P, Bernard S. Ketamine as an analgesic in the pre-hospital setting: a systematic review. Acta Anaesthesiol Scand. 2011 Jul;55(6):638-43. doi: 10.1111/j.1399-6576.2011.02446.x. Epub 2011 May 16. PMID 21574967
- [Background] Green SM, Andolfatto G, Krauss BS. Ketamine and intracranial pressure: no contraindication except hydrocephalus. Ann Emerg Med. 2015 Jan;65(1):52-4. doi: 10.1016/j.annemergmed.2014.08.025. Epub 2014 Sep 20. No abstract available. PMID 25245275
- [Background] Graudins A, Meek R, Egerton-Warburton D, Oakley E, Seith R. The PICHFORK (Pain in Children Fentanyl or Ketamine) trial: a randomized controlled trial comparing intranasal ketamine and fentanyl for the relief of moderate to severe pain in children with limb injuries. Ann Emerg Med. 2015 Mar;65(3):248-254.e1. doi: 10.1016/j.annemergmed.2014.09.024. Epub 2014 Nov 18. PMID 25447557
- [Background] Woolf CJ. Central sensitization: implications for the diagnosis and treatment of pain. Pain. 2011 Mar;152(3 Suppl):S2-S15. doi: 10.1016/j.pain.2010.09.030. Epub 2010 Oct 18. PMID 20961685
- [Background] Kulbe J. The use of ketamine nasal spray for short-term analgesia. Home Healthc Nurse. 1998 Jun;16(6):367-70. No abstract available. PMID 9708149
- [Background] Plunkett A, Turabi A, Wilkinson I. Battlefield analgesia: a brief review of current trends and concepts in the treatment of pain in US military casualties from the conflicts in Iraq and Afghanistan. Pain Manag. 2012 May;2(3):231-8. doi: 10.2217/pmt.12.18. PMID 24654665
- [Background] Reid C, Hatton R, Middleton P. Case report: prehospital use of intranasal ketamine for paediatric burn injury. Emerg Med J. 2011 Apr;28(4):328-9. doi: 10.1136/emj.2010.092825. Epub 2011 Feb 3. PMID 21292791
- [Background] Andolfatto G, Willman E, Joo D, Miller P, Wong WB, Koehn M, Dobson R, Angus E, Moadebi S. Intranasal ketamine for analgesia in the emergency department: a prospective observational series. Acad Emerg Med. 2013 Oct;20(10):1050-4. doi: 10.1111/acem.12229. PMID 24127709
- [Background] Carr DB, Goudas LC, Denman WT, Brookoff D, Staats PS, Brennen L, Green G, Albin R, Hamilton D, Rogers MC, Firestone L, Lavin PT, Mermelstein F. Safety and efficacy of intranasal ketamine for the treatment of breakthrough pain in patients with chronic pain: a randomized, double-blind, placebo-controlled, crossover study. Pain. 2004 Mar;108(1-2):17-27. doi: 10.1016/j.pain.2003.07.001. PMID 15109503
- [Background] Galinski M, Dolveck F, Combes X, Limoges V, Smail N, Pommier V, Templier F, Catineau J, Lapostolle F, Adnet F. Management of severe acute pain in emergency settings: ketamine reduces morphine consumption. Am J Emerg Med. 2007 May;25(4):385-90. doi: 10.1016/j.ajem.2006.11.016. PMID 17499654
- [Background] Marland S, Ellerton J, Andolfatto G, Strapazzon G, Thomassen O, Brandner B, Weatherall A, Paal P. Ketamine: use in anesthesia. CNS Neurosci Ther. 2013 Jun;19(6):381-9. doi: 10.1111/cns.12072. Epub 2013 Mar 22. PMID 23521979
- [Background] Malinovsky JM, Servin F, Cozian A, Lepage JY, Pinaud M. Ketamine and norketamine plasma concentrations after i.v., nasal and rectal administration in children. Br J Anaesth. 1996 Aug;77(2):203-7. doi: 10.1093/bja/77.2.203. PMID 8881626
- [Background] Yanagihara Y, Ohtani M, Kariya S, Uchino K, Hiraishi T, Ashizawa N, Aoyama T, Yamamura Y, Yamada Y, Iga T. Plasma concentration profiles of ketamine and norketamine after administration of various ketamine preparations to healthy Japanese volunteers. Biopharm Drug Dispos. 2003 Jan;24(1):37-43. doi: 10.1002/bdd.336. PMID 12516077
- [Background] Weber F, Wulf H, Gruber M, Biallas R. S-ketamine and s-norketamine plasma concentrations after nasal and i.v. administration in anesthetized children. Paediatr Anaesth. 2004 Dec;14(12):983-8. doi: 10.1111/j.1460-9592.2004.01358.x. PMID 15601346
- [Background] Huge V, Lauchart M, Magerl W, Schelling G, Beyer A, Thieme D, Azad SC. Effects of low-dose intranasal (S)-ketamine in patients with neuropathic pain. Eur J Pain. 2010 Apr;14(4):387-94. doi: 10.1016/j.ejpain.2009.08.002. Epub 2009 Sep 3. PMID 19733106
- [Background] Yeaman F, Meek R, Egerton-Warburton D, Rosengarten P, Graudins A. Sub-dissociative-dose intranasal ketamine for moderate to severe pain in adult emergency department patients. Emerg Med Australas. 2014 Jun;26(3):237-42. doi: 10.1111/1742-6723.12173. Epub 2014 Apr 8. PMID 24712757
- [Background] Jensen MP, Martin SA, Cheung R. The meaning of pain relief in a clinical trial. J Pain. 2005 Jun;6(6):400-6. doi: 10.1016/j.jpain.2005.01.360. PMID 15943962
- [Background] Ferreira-Valente MA, Pais-Ribeiro JL, Jensen MP. Validity of four pain intensity rating scales. Pain. 2011 Oct;152(10):2399-2404. doi: 10.1016/j.pain.2011.07.005. PMID 21856077
- [Background] Bahreini M, Jalili M, Moradi-Lakeh M. A comparison of three self-report pain scales in adults with acute pain. J Emerg Med. 2015 Jan;48(1):10-8. doi: 10.1016/j.jemermed.2014.07.039. Epub 2014 Sep 27. PMID 25271179
- [Derived] Andolfatto G, Innes K, Dick W, Jenneson S, Willman E, Stenstrom R, Zed PJ, Benoit G. Prehospital Analgesia With Intranasal Ketamine (PAIN-K): A Randomized Double-Blind Trial in Adults. Ann Emerg Med. 2019 Aug;74(2):241-250. doi: 10.1016/j.annemergmed.2019.01.048. Epub 2019 Mar 27. PMID 30926189
- See also: British Columbia Ambulance Service information page. — http://www.bcehs.ca/our-services/programs-services/ground-ambulances